CLINICAL TRIAL: NCT06328166
Title: The Effect and Safety of Recombinant Human Fibroblast Growth Factor-1 for Patient With Carpal Tunnel Syndrome
Brief Title: The Effect and Safety of Recombinant Fibroblast Growth Factor-1 for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: Eusol Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yu-CHI Su, Attending Physician and lecturer of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rFGF-1 for CTS
Record Dates: First submitted 2023-12-03; First posted 2024-03-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; recombinant human fibroblast growth factor 1
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- recombinant human fibroblast growth factor 1 (ES135) (Experimental): Ultrasound-guided injection with recombinant human fibroblast growth factor 1 (ES135) between carpal tunnel and median nerve.
  Interventions: Procedure: Sono-guided injection with ES135
- normal saline (Placebo Comparator): Ultrasound-guided injection with normal saline between carpal tunnel and median nerve.
  Interventions: Procedure: Sono-guided injection with placebo

INTERVENTIONS:
Procedure: Sono-guided injection with ES135 — Sono-guided injection with ES135 between carpal tunnel and median nerve
  Arms: recombinant human fibroblast growth factor 1 (ES135)
Procedure: Sono-guided injection with placebo — Sono-guided injection with placebo between carpal tunnel and median nerve
  Arms: normal saline

SUMMARY:
Carpal tunnel syndrome (CTS) is a common peripheral entrapment mononeuropathy of the upper limb, which results from compression of median nerve at level of wrist. In recent years, regenerative medicine has gradually been applied in the treatment of various degenerative conditions such as bones, muscles, and nerves. Human fibroblast growth factor 1 is a single-chain protein , which has been shown to play a crucial regulatory role in the brain and spinal cord and can facilitate nerve cell differentiation and growth. ES135 is a recombinant human fibroblast growth factor 1 (rhFGF1) which is composed of 135 amino acids with a molecular weight of approximately 15.2 kilodalton. Several studies have shown that significant improvement of Functional Independence Measure, motor and sensory function of spinal cord injury patients after ES135 treatment. One study also revealed the muscle strength have significant improvement in brachial plexus injury patients after ES135 therapy. According to above studies, the investigators hypothesized that ES135 may have benefits to CTS patients. Hence, the purpose of this study aim to demonstrate the therapeutic effects and safety of ES135 for CTS.

DETAILED DESCRIPTION:
Participants established with diagnosis of mild-to-moderate CTS will been randomly assigned to ES135 or Placebo groups. With ultrasound guidance, injection with ES135 or Placebo was performed between median nerve and transcarpal ligament. The Boston Carpal Tunnel Syndrome Questionnaire is assigned as primary outcome. The secondary outcomes encompass visual analog scale, electrophysiological studies and cross-sectional area of the median nerve. The assessment is performed prior injection and at 1, 2, 3, 4 and 6 months post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 year-old.
* Diagnosis was confirmed by using an electrophysiological study
* CTS symptoms for more than 3 months.

Exclusion Criteria:

* Severe CTS
* Allergy to ES135
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid/platelet-rich plasma injection for CTS within 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 1st month, 2nd month, 3rd month,4th month, 6th month after injection. | Pre-treatment, 1st month, 2nd month, 3rd month,4th month, 6th month.
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 1st month, 2nd month, 3rd month,4th month, 6th month after injection. | Pre-treatment, 1st month, 2nd month, 3rd month,4th month, 6th month.
  Digital pain severity or paresthesia/dysesthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 1st month, 2nd month, 3rd month,4th month, 6th month after injection. | Pre-treatment, 1st month, 2nd month, 3rd month,4th month, 6th month.
  Using the musculoskeletal sonogram to measure the cross-sectional area (mm2) of the median nerve before treatment and multiple time frame after treatment
Change from baseline of conduction velocity, latency of median nerve on 1st month, 2nd month, 3rd month,4th month, 6th month. | Pre-treatment, 1st month, 2nd month, 3rd month,4th month, 6th month.
  electrophysiological study of the median nerve: Distal motor latency (ms)、Sensory nerve conduction velocity (m/s) before treatment and multiple time frame after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Tri-Service General Hospital, School of Medicine, National Defense Medical Center; Yu Chi Su, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- No. 325, Sec. 2, Chenggong Rd., Neihu Dist., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254
- [Background] Javerzat S, Auguste P, Bikfalvi A. The role of fibroblast growth factors in vascular development. Trends Mol Med. 2002 Oct;8(10):483-9. doi: 10.1016/s1471-4914(02)02394-8. PMID 12383771
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Huang GS, Chen LC. Six-month efficacy of platelet-rich plasma for carpal tunnel syndrome: A prospective randomized, single-blind controlled trial. Sci Rep. 2017 Dec;7(1):94. doi: 10.1038/s41598-017-00224-6. Epub 2017 Mar 7. PMID 28273894
- [Background] Wu JC, Huang WC, Huang MC, Tsai YA, Chen YC, Shih YH, Cheng H. A novel strategy for repairing preganglionic cervical root avulsion in brachial plexus injury by sural nerve grafting. J Neurosurg. 2009 Apr;110(4):775-85. doi: 10.3171/2008.8.JNS08328. PMID 19119881
- [Background] Teng YD, Mocchetti I, Wrathall JR. Basic and acidic fibroblast growth factors protect spinal motor neurones in vivo after experimental spinal cord injury. Eur J Neurosci. 1998 Feb;10(2):798-802. doi: 10.1046/j.1460-9568.1998.00100.x. PMID 9749747
- [Background] Wu JC, Huang WC, Chen YC, Tu TH, Tsai YA, Huang SF, Huang HC, Cheng H. Acidic fibroblast growth factor for repair of human spinal cord injury: a clinical trial. J Neurosurg Spine. 2011 Sep;15(3):216-27. doi: 10.3171/2011.4.SPINE10404. Epub 2011 Jun 10. PMID 21663406